CLINICAL TRIAL: NCT00749229
Title: Prospective Cohort Study on the Feasibility and Reliability of 'Open' Balloon Kyphoplasty in Types A3.2, A3.3, B1 and C1 MAGERL Classification Vertebral Fractures(STIC 4)
Brief Title: Feasibility Study of Balloon Kyphoplasty in Traumatic Vertebral Fractures Needing Surgical Fixation
Acronym: TRAUMAA3B1C1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the number of patients recruited at present is sufficient for analysis.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P060109
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2014-12

CONDITIONS: One or Two Traumatic Vertebral Fractures; Located Between T11 and L5; Balloon Kyphoplasty
Keywords: Traumatic vertebral fracture; Balloon Kyphoplasty; type A3.2, or A3.3 or B1 or C1 in the MAGERL CLASSIFICATION
MeSH Terms: interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Balloon kyphoplasty
  Interventions: Device: balloon kyphoplasty

INTERVENTIONS:
Device: balloon kyphoplasty — During the same surgery or some days later on, percutaneous Balloon kyphoplasty of the fractured vertebral body (ies) using polymethylmetacrylate cement injection through a posterior transpedicular approach will be carried out in replacement of anterior spine surgery to restore vertebral body strength

SUMMARY:
Some unstable traumatic vertebral fractures (types A3.2, A3.3, B1 et C1 according to MAGERL classification) may undergo unpredictable secondary displacement. Such fractures require a two session surgery with a first operation carried out immediately to achieve posterior fixation and a second surgery which is performed some days later to stabilize the anterior spine and restore stress resistance.

Goal of the present study is to show that percutaneous Balloon Kyphoplasty is able to restore anterior spine strength and replace second session surgery.

DETAILED DESCRIPTION:
Patients with traumatic vertebral fractures type A3.2, A3.3, B1 and C1 of the MAGERL classification will be enrolled in this open study. They will be operated on in emergency to perform spinal canal decompression, fracture reduction and posterior fixation using fixation plates with pedicular screws combined with bone graft.

During the same surgery or some days later on, percutaneous Balloon kyphoplasty of the fractured vertebral body (ies) using polymethylmetacrylate cement injection through a posterior transpedicular approach will be carried out in replacement of anterior spine surgery to restore vertebral body strength.Patients will be followed up for one year.

Expected advantages of this management compared the conventional two session surgery include the following:

* decreased morbidity due to suppression of the anterior surgery
* improve final spine alignment and vertebral Kyphotic angle avoiding the loss in kyphotic angle which often occurs between the posterior and anterior surgery with the conventional two session surgery.

ELIGIBILITY:
Inclusion Criteria:

* Preliminary clinical examination (the anaesthesist must have provided his approval for the surgical procedure)
* Patient must have signed the consent form
* Male or female patient aged 18 or over
* One or two traumatic vertebral fractures located between T11 and L5 and type A3.2, A3.3, B1 or C1 in the MAGERL classification, and with a regional kyphotic angle > 15° and treated by osteosynthesis through a posterior surgical approach with or without spinal decompression
* Fracture with or without neurological difficulties
* Non tumoral origin: Confirmed by biopsy at the same time of the Balloon Kyphoplasty procedure.

Exclusion Criteria:

* Non- traumatic, malignant or osteoporotic vertebral fractures
* History of surgical or percutaneous spine treatment except simple discectomy at a single or multiple vertebral levels with no residual pain.
* Known allergy to a contrast media or to one of the cement components used for kyphoplasty.
* More than two recent vertebral fractures
* Current infection
* Impossibility to perform the percutaneous approach of the vertebra to treat.
* Reduction by more than 50% of the anteroposterior width of the bony spinal canal due to the vertebral fracture to treat.
* Vertebral fracture with loss of 90%or more of the vertebral body height
* Patient presenting a non correctable spontaneous or therapeutic coagulation disorder.
* Evolutive cardiac disease nonreactive to medical treatment
* Non compliant patient: Impossibility to participate to the study and to be followed up for 1 year.
* Pregnant or breast feeding women
* Patient not affiliated to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Loss of less than 10 degrees in spine kyphosis angle at one year follow-up after surgery compared to postoperative measurements | 1 year

SECONDARY OUTCOMES:
Pain evaluation using a visual analogic scale | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
EIFEL questionnaire for back pain evaluation | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Quality of life evaluation (SF 12). | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Analgesics intake according to the WHO classification (Classes 1, 2 and 3). | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Regional spine Kyphosis angle and global thoracic and lumbar Kyphosis angle. | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Changes in anterior, mid and posterior vertebral heights of the treated vertebral body | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Changes in height of the intervertebral disc spaces adjacent to the treated vertebra. | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Number of new vertebral fractures occurring during the one year follow-up period. | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Cost evaluation in a sample of 10% of patients randomly selected including the following costs : o Intervention cost.o Medical treatment costs o Consultation costs. o Hospitalization cost o Complication costs | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Follow-up of anterior, median and posterior height of the treated vertebral body, obtained by making an average of all measurements, on 3 cuts tomodensitometry (TDM) on the sagittal level : lateral right, median and lateral left | preoperative, at J6 and at J360

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis LAREDO, M.D.,PR., Principal Investigator — AP/HP Assistance Publique-Hôpitaux de Paris
Locations (1):
- Service de Radiologie, Hôpital Lariboisière, Paris, France